CLINICAL TRIAL: NCT05353231
Title: Brief Mental Training and Internal Attentional Control in Repetitive Negative Thinking: Experimental Laboratory Investigation
Brief Title: Brief Mental Training and Internal Attentional Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MDTT-AFACT
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Attention Impaired; Mental Health Issue; Rumination
Keywords: Cognitive Change; Internal attention; Interoceptive attention; Meditation; Mindfulness; Computerized intervention; Attentional bias
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 - Attention Feedback Awareness and Control Training (Experimental)
  Interventions: Behavioral: Attention Feedback Awareness and Control Training (A-FACT)
- Intervention 2 - Mindful Disengagement from Thoughts Training (Experimental)
  Interventions: Behavioral: Mindful Disengagement from Thoughts Training (MDTT)
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo-Control

INTERVENTIONS:
Behavioral: Attention Feedback Awareness and Control Training (A-FACT) — A-FACT is designed to promote meta-awareness of moment-to-moment biased internal attention allocation (e.g. toward negative thoughts) and thereby internal attentional control.
  Participants will be instructed that they will complete a task designed to reduce their attentional bias to some thoughts. Following a fixation que, the auditory neutral or negative simulated thought stimulus is delivered, and 500ms prior to termination of the auditory stimulus, a visual stimulus is presented until participants categorize the visual stimulus as greater than or smaller than 5 objects. Latency to disengage attention from each thought stimuli, at the trial-level, is repeatedly measured, and after each negative thought stimulus, trial-level feedback on the latency to disengage is delivered back to participants through a visual scale representing their attentional bias. Participants will complete approximately 100 trials in total wherein randomly 1 or 2 neutral trials follow each negative trial.
  Arms: Intervention 1 - Attention Feedback Awareness and Control Training
Behavioral: Mindful Disengagement from Thoughts Training (MDTT) — MDTT is designed to promote meta-awareness of moment-to-moment biased internal attention allocation (e.g. toward negative thoughts) and thereby internal attentional control. Participants will be instructed that they will complete a task designed to reduce their attentional bias to some thoughts. Participants will first learn and practice a focused attention on the breath meditation. Then, participants will practice pressing a button each time they notice an inhalation or exhalation during the focused attention meditation. Next, during the meditation, participants will be presented the auditory neutral or negative simulated thought stimuli and will train internal attentional control by repeatedly disengaging their attention from these stimuli and back to their breath MDTT will thus entail 80 trials (40 negative, 40 neutral, ITI ≈ 10sec) during the focused attention on the breath meditation.
  Arms: Intervention 2 - Mindful Disengagement from Thoughts Training
Behavioral: Placebo-Control — The condition is designed as a placebo control for the Attention Feedback Awareness and Control Training (A-FACT) training condition. Participants will be instructed that they will complete a task designed to reduce their attentional bias to some thoughts. Rather than the quantity categorization task with trial-level feedback, participants only engage in the quantity categorization task. The task is identical in all other ways to the A-FACT condition. Participants will complete approximately 100 trials in total wherein randomly 1 or 2 neutral trials follow each negative trial.
  Arms: Placebo

SUMMARY:
Previous research documented that real-time feedback on attention as well as related forms of mental training (e.g. mindfulness meditation) may be used to train and impact external attentional control. These approaches to mental training are designed to train meta-awareness in order to enable attentional control. It is not yet known, however, whether such training targeting meta-awareness can be similarly used to impact internal attentional control. Thus, the investigators will test whether real-time feedback training and a brief mindfulness meditation training, relative to placebo control, will lead to greater internal attentional control among adults with elevated negative repetitive thinking.

DETAILED DESCRIPTION:
Participants will complete all assessments and training in a single laboratory session. Participants (N=105) with elevated levels of negative repetitive thinking (Rumination Response Scale -Brooding >=11) will be randomly assigned to one of 3 intervention arms: Attention Feedback Awareness and Control Training (A-FACT; n=35), Mindful Disengagement from Thoughts Training (MDTT; n=35), or placebo control (n=35).

At pre- and post-intervention, the investigators will measure: (1) Subjective emotional reactivity in response to negative vs. neutral self-referential thoughts using the Simulated Thought Paradigm (STP)-Emotional Reactivity task; (2) Interoceptive attention (i.e. sensibility) of the subjective location, intensity and hedonic tone of bodily sensations, using the STP-Body Map task, and (3) internal attentional control (i.e. latency to disengage) using the STP-Digit Categorization Task.

At post-intervention assessment only, the investigators will measure: (1) Meta-awareness of internal attentional dyscontrol using the STP-Digit Categorization Task with Self-Caught Probes; (2) internal attentional control (i.e. selective attention) using the STP-One-Back Dichotic Listening Task as a measure of the generalizability of the expected primary effect on internal attentional control.

The primary aim is to test the effect of 2 active intervention arms, Attention Feedback Awareness and Control Training and Mindful Disengagement from Thoughts Training, relative to one another and placebo control, on internal attentional control from pre-to-post training among adults with elevated negative repetitive thinking. The investigators hypothesise that both active interventions conditions will yield improvement in internal attentional control, as measured by the Digit Categorization Task integrated with the Simulated Thoughts Paradigm, from pre-to-post intervention, relative to the placebo-control.

Secondary aims are to test the effects of the 2 active intervention arms, relative to one another and placebo control, on subjective emotional reactivity to negative self-referential thoughts, selection bias to negative self-referential thoughts, meta-awareness of attentional dyscontrol, as well as interoceptive attention to bodily sensations in response to negative self-referential thoughts. The investigators hypothesize that, relative to the control-placebo group, the active intervention groups will yield (a) reduced emotional reactivity to negative self-referential thoughts as measured in the Emotional Reactivity Task, (b) higher levels of meta-awareness of attentional dyscontrol as measured by the STP-Digit Categorization Task with Self-Caught Probes, and (c) higher levels of selective internal attentional control as measured by the STP-One-Back Dichotic Listening Task.

Additionally, the investigators hypothesize that, relative to the placebo control group and the Attention Feedback Awareness and Control Training group, the Mindful Disengagement from Thoughts Training group will yield enhanced interoceptive attention (i.e. sensibility) to a broader range of locations (e.g. peripheral body areas), intensities (e.g. subtle sensations) and hedonic tones (e.g. neutral and pleasant hedonic tones) of bodily sensations in response to self-referential thoughts, as measured by STP-Body Map task.

Finally, the investigators hypothesized non-inferiority between the active intervention groups with respect to all mentioned measured outcomes, with exception of the noted STP-Body-Map Task.

ELIGIBILITY:
Inclusion Criteria:

* Brooding subscale in the Ruminative Responses Scale (RRS) - with score equal to or greater than 11

Exclusion Criteria:

* Endorsement of suicidal ideation ("Yes" answer to Patient Health Questionnaire - 9 Item
* Psychotic Symptoms, specifically auditory hallucinations
* Self-report lack of fluency in speaking or understanding Hebrew-language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the STP-Digit Categorization Task | pre-intervention, immediately post-intervention
  The STP-Digit Categorization Task (STP-DCT) will be used to measure change, from pre-intervention to post-intervention, in internal attentional disengagement. Attentional disengagement will be computed by the difference in reaction time on negative relative to neutral simulated thought stimuli as well as via a dynamic bias score calculated by subtracting the running mean of the 8 neutral trials window ( 4 neutral trials backwards and 4 neutral trials forward), from each negative trial reaction time that exceeds the 95%CI., dividing this distance by the 8 neutral trials window standard deviation (Amir, Ruimi, & Bernstein, 2021). A positive score reflects greater difficulty to disengage from negative relative to neutral thought stimuli.

SECONDARY OUTCOMES:
STP-One-Back Dichotic Listening Task | immediately post-intervention
  The STP-One-Back Dichotic Listening Task will be used to measure biased selective attention of negative simulated thought stimuli. Biased selective attention will be computed by the difference in accuracy for negative relative to neutral simulated thought stimuli. An accurate response (for each stimulus) is the correct left/right button press for the respective left/right channel in which a repetition of auditory neutral or negative simulated thought stimuli were presented - i.e., the stimulus delivered at trial n-1 was repeated on trial n (in the same channel); or the correct withholding of a response if no repetition was present. A positive bias score reflects greater selective attention to negative relative to neutral thought stimuli.
STP-Digit Categorization Task (STP-DCT) with Self-Caught Probes | immediately post-intervention
  The STP-Digit Categorization Task (STP-DCT) with Self-Caught Probes will be used to measure meta-awareness of attentional disengagement from stimulated thoughts stimuli. While performing the STP-DCT task, participants are instructed to, on the trial-level, report when the simulated thought influenced their trial response (i.e., led to difficulty disengaging attention from thought to categorize the digit) by pressing a key immediately following trial response. Meta-awareness will be computed using the Diagnostic Odds Ratio (Ruimi, Hadash, Zvielli, Amir, Goldstein, & Bernstein, 2018). Positive scores reflects degree of meta-awareness for difficulty to disengage from thought stimuli.
Change in the STP-Emotional Reactivity Task | pre-intervention, immediately post-intervention
  The STP-Emotional Reactivity Task will be used to measure change, from pre- to post-intervention, in emotional reactivity to negative simulated thought stimuli. Emotional reactivity will be computed as the difference between the mean of 5 subjective emotion stats (irritability, anger, anxiety, guilt, distress), each self-rated on a 5-point Likert-type scale, following one block of 20 neutral-, and then again one block of 20 negative- simulated thought stimuli. Positive scores reflect greater emotional reactivity in response to negative relative to neutral thought stimuli.
Change in the STP-Body Map Task | pre-intervention, immediately post-intervention
  The STP-Body Map Task will be used to measure interoceptive attention via subjective assessment (i.e. sensibility) of bodily sensations, following negative and neutral stimuli (STP). The following interoceptive attention variables will be calculated: (1) Detection of bodily sensations (frequency (number) of bodily sensations); (2) Magnitude of bodily sensations (mean intensity of bodily (range from 1 to 5)); (3) Bias to hedonic tone of bodily sensations (proportion/percent of neutral, pleasant and unpleasant sensations), (4) Bias to central vs peripheral bodily sensations (e.g. proportion/percent of sensations in torso/head vs. legs/arms).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bernstein, Ph.D., Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code